CLINICAL TRIAL: NCT01773252
Title: A With-in Subject, Controlled Study to Determine the Sensitivity and Specificity of the Cardiox Flow Detection System for the Detection of Right-to-Left Cardiac Shunts Compared to Transesophageal Echocardiography and Transcranial Doppler Ultrasound
Brief Title: Right to Left Cardiac Shunt Detection
Acronym: PFO Detection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to perform a market withdrawal of the product
Sponsor: Cardiox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FDS-0005
Record Dates: First submitted 2013-01-08; First posted 2013-01-23 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Right to Left Shunt; Patent Foramen Ovale; Atrial Septal Defect
Keywords: RLS; RTLS; PFO; ASD; shunt; cardiac; paradoxical thromboembolism; interventional cardiology; stroke; migraine; aura; obstructive sleep apnea; decompression illness; neurology; transesophageal echocardiography; TEE; transthoracic echocardiography; TTE; transcranial Doppler; ultrasound; TCD; power m Mode; indocyanine green dye; ICG; Valsalva
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Septal Defects, Atrial; Stroke; Migraine Disorders; Epilepsy; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEE (Experimental): Within patient comparison of TEE, FDS and a TCD from select study sites
  Interventions: Device: Flow Detection System

INTERVENTIONS:
Device: Flow Detection System
  Other Names: Model 100

SUMMARY:
The purpose of this study is to evaluate the sensitivity and specificity of the Cardiox Flow Detection System (FDS) in identifying an intracardiac right-to-left shunt (RLS) compared to the results of transesophageal echocardiography (TEE).

RLS intracardiac shunts are associated with a number of clinically important syndromes including paradoxical thromboembolism (causing stroke or other systemic infarct), migraine headaches (particularly with aura), desaturation with obstructive sleep apnea, and decompression illness. From a research perspective, the detection of shunts in subjects with these types of syndromes is critical in helping to define the role of RLS in these disease processes. From a clinical perspective, shunt detection will be increasingly important in an era where interventional procedures for repairing cardiac defects are available for subjects determined to be at risk.

The currently accepted reference standard for detection of an intra-cardiac patent foramen ovale/atrial septal defect (PFO/ASD) RLS is a transesophageal echocardiography (TEE), a procedure that is invasive, uncomfortable, and requires conscious sedation.

Alternative options include transthoracic echocardiography (TTE) with injection of agitated saline (with and without Valsalva strain), a procedure that is far less sensitive than TEE due to the echocardiography imaging limitations seen in many adults.

Finally, transcranial Doppler (TCD) with injection of agitated saline (with and without Valsalva strain) is a newer entrant into this arena that does not require sedation or any invasive instrumentation.

The Cardiox Model 100 FDS utilizes an optical sensor positioned on the surface of the subject's skin at the scaphoid fossa of the ear. Next, a predetermined dose of an indicator dye, indocyanine green (ICG), is injected at a predetermined rate into a peripheral antecubital vein of the subject while the subject performs a breathing maneuver called a Valsalva maneuver. The exhalation by the subject into a mouthpiece connected to a pressure transducer via a flexible tubing extension, or its equivalent (ie, performing the Valsalva maneuver), is an essential step for all existing RLS detection methods. The Valsalva maneuver by the subject creates a pressure differential between the right and left sides of the heart. This Valsalva maneuver results in blood flow from the right side of the heart to the left side of the heart through an ASD, and/or causes a PFO, if present, to open, also allowing blood to flow directly from the right side to the left side of the heart without passing through the lungs (pulmonary vasculature) for oxygenation.

The Earpads, including their fluorescence sensor arrays (FSA), are used to measure the relative concentration (ie, fluorescence signal level) of ICG dye in the bloodstream as a function of time. If a premature inflection or peak occurs in the ICG dye concentration level at a time point prior to the rise and fall of the concentration associated with the main bolus of indicator, then a RLS is present in the heart. The amplitude of this premature ICG dye-dilution curve (referred to as "RLS-indicator dilution curve") is used to subsequently quantify the magnitude of the right-to-left shunt by ratiometrically comparing the amplitude of this RLS indicator dilution curve to the amplitude of the main indicator dilution curve associated with that portion of the injected ICG dye that follows the normal pathway from the right side of the heart, through the lungs, and into the left side of the heart (referred to as "normal indicator dilution curve").

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Is currently scheduled (within five days of FDS) for a TEE study with agitated saline contrast (bubble study) or has had a TEE procedure with agitated saline contrast study (bubble study) within the previous 12 months;
* If the Subject has undergone a shunt closure procedure, the protocol related TEE must be conducted greater than 12 months post closure.
* Is able to read and understand the ICF and has voluntarily provided written informed consent;
* Subject is able to perform a successful Valsalva maneuver (obtaining a score of 3 stars) using the Cardiox FDS device.

Exclusion Criteria:

* Subjects with known allergy or sensitivity to ICG or to iodide contrast dye or iodides including medications with high iodine content;
* Pregnant women or nursing mothers;
* Subjects scheduled for a radioactive iodine uptake studies (eg, thyroid studies) within one week of completing this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Presence or absence of shunt | Five days
  To establish the sensitivity and specificity of the Cardiox FDS using transesophageal echocardiography (TEE) as the reference standard
Adverse Events | Five days
  To establish the safety of the Cardiox FDS device

SECONDARY OUTCOMES:
Presence or absence of shunt | Three days
  To establish the positive percent agreement and the negative percent agreement of Cardiox FDS procedure with a transcranial Doppler (TCD) from select study sites.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Jopling, MD, Study Director — Cardiox Corporation
Locations (8):
- United States (8):
  - Heart and Vascular Center of Arizona, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Methodist DeBakey Heart and Vascular Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington